CLINICAL TRIAL: NCT05448612
Title: Comparative Effect of Active Release Technique and Muscles Energy Technique on Pain, ROM and Functional Disability in Adhesive Capsulitis Patients With Trigger Points
Brief Title: Comparative Effect of ART and MET on Pain, ROM and Functional Disability in AC Patients With Trigger Points
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-/98-04/2022
Record Dates: First submitted 2022-05-22; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-05

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive capsulitis; Trigger points; Active release technique; Muscle energy technique
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Release Technique (Experimental): In ART the particular muscle is taken from shortened to lengthened position or vice versa. Duration of treatment will be of 8-15min
  Interventions: Other: Active Release Technique and muscle energy technique
- Muscles Energy Technique (Experimental): In METs,the protocol will perform for 3 repetitions per day and thrice a week for 5 week.
  Interventions: Other: Active Release Technique and muscle energy technique

INTERVENTIONS:
Other: Active Release Technique and muscle energy technique — 74 participants divided into two groups and 37 in each group.

SUMMARY:
The aim of this study to determine the Comparative effect of active release technique and muscle energy technique on pain, ROM and functional disability in adhesive capsulitis patients with trigger points.

DETAILED DESCRIPTION:
74 participants are included in this study in two groups and 37 for each group. Group A for active release technique along with conventional therapy and Group B for muscles energy technique along with conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female.
* Participants having unilateral adhesive capsulitis.
* Participants with sub-acute adhesive capsulitis.
* Participants having age of 40-60 years.

Exclusion Criteria:

* Patient with cervical radiculopathy.
* Fractures of upper limb.
* Thoracic outlet syndrome.
* Post-traumatic.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Numerical pain rating scale | Change from Baseline in pain to 6 week
  patients rate their pain from 0 to 10, from 0 to 20, or from 0 to 100. Zero represents "no pain," whereas 10, 20, or 100 represents the opposite end of the pain continuum (e.g., "the most intense pain imaginable," "pain as intense as it could be," "maximum pain").
Universal Goniometry | Change from Baseline in range of motion to 6 week
  Universal goniometer (UG) is commonly used as a standard method to evaluate range of motion (ROM) as part of joint motions.
Shoulder Pain and Functional Disability Index | Change from Baseline in disability to 6 week
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire consisting of items grouped into pain and disability subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Shahzadi Sumbal Naz, Dpt, Study Chair — UOL
Locations (1):
- Spot Rehab, Lahore, Pakistan